CLINICAL TRIAL: NCT02375321
Title: Quality of Life in Patients With Obstructive Sleep Apnea: The Role of CPAP Associated to Psychological Support
Acronym: QUOLOSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Careggi Hospital (Other)
Responsible Party: Principal Investigator, Corrado Antonio, M. D, Chief of Respiratory Intensive Care Unit, MD, Careggi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rubrica n. SPE 14.015
Record Dates: First submitted 2015-02-18; First posted 2015-03-02 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Obstructive Sleep Apnea; Depressive Symptoms
Keywords: OSA; Depression; Quality of Life; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Study Group: patients with OSA and depressive symptoms treated with CPAP and psychological support
  Interventions: Behavioral: CPAP and Psychological support
- Group B (No Intervention): Control Group: patients with OSA and depressive symptoms treated with CPAP

INTERVENTIONS:
Behavioral: CPAP and Psychological support — Six sessions of psychological support with cognitive behavioural orientation lasting 1 hour every two weeks for 3 months
  Arms: Group A

SUMMARY:
Many researches have shown that patients with Obstructive Sleep Apnea (OSA) and often also the family members have a decreased quality of life, problems related to the sexual sphere, depressive disorders and anxiety problems. To date still remains controversial the relationship between OSA and quality of life, also the link between sleep apnea syndrome and depression is unclear.

In adult patients with OSA the treatment of choice is the application of a continuous positive airway pressure (CPAP: Continuous Positive Airway Pressure) at the opening of the airways. With the CPAP treatment the sleep normalizes and daytime sleepiness fades or disappears.

Many studies have shown that this treatment determines improvement of the medical and psychological status. However, the rate of non-adherence to treatment reported in the literature is about 46-83%, considering as adherence the use of CPAP for at least 4 hours per night. A recent study has shown that CPAP used as a single treatment in patients with OSA and depression, has reduced the depressive symptoms but in a significant percentage of patients (42%), the depressive symptoms remained unchanged or worsened. At the present time have not been published, to our knowledge, studies concerning the effectiveness of the combined treatment of CPAP and psychological support on the mood and on the quality of life OSA patients.

Therefore the aim of this study is to evaluate the effects of the combined treatment with CPAP and psychological intervention with cognitive behavioural therapy on the mood and on the quality of life of OSA patients.

DETAILED DESCRIPTION:
Primary endpoint The primary endpoint of the study is the evaluation of the mood tone, measured before and 12 weeks after the start of treatment through the administration of the13-item self-rated Pichot depression scale (QD2A). Each subject will be assigned to one of the following categories:"absence of alterations in mood" or "presence of mood disorders," according to the test result (score <7 or score ≥7).

The subjects in which, for whatever reason, the QD2A test after 12 weeks of treatment will not be available, will be considered failures, and will be assigned to the class "presence of mood disorders." Secondary endpoint Evaluation of adherence to CPAP treatment, considering as adherence the use of CPAP, during the observation period, for at least 4 hours per night.

After 12 weeks of treatment, each patient will be classified as "adherent" or "non-adherent" to the treatment itself. The subjects in whom, for whatever reason, after 12 weeks of treatment, the total number of hours of use of CPAP will not be available, will be assigned to the class of "non-adherent".

ELIGIBILITY:
Inclusion Criteria:

* all patients with a known diagnosis of obstructive sleep apnea who need of treatment with CPAP
* aged 18-70 years
* presence of alteration of mood, identified by a score of ≥7 by means the QD2A test
* written informed consent, signed and dated

Exclusion Criteria:

* previous treatment for OSA
* sleep disorders different from OSA
* cognitive impairment diseases
* severe psychiatric disorders
* alcoholism or other abuses.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
The difference between the proportion of subjects with no alterations of mood, measured by means of the QD2A test, before and 12 weeks after the start of treatment, observed in the CPAP group plus psychological support and only CPAP treatment | 3 months

SECONDARY OUTCOMES:
The difference between the proportion of subjects adherent to CPAP treatment in both groups, considering as adherence the use of CPAP, during the observation period, for at least 4 hours per night. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Corrado, MD, Principal Investigator
Locations (1):
- Careggi Hospital - Terapia Intensiva Pneumologica, Florence, Fi, Italy

REFERENCES:
- [Background] Sampaioa R, Pereira MG, Winck JC. Psychological morbidity, illness representations, and quality of life in female and male patients with obstructive sleep apnea syndrome. Psychology, Health & Medicine 2 (17): 136-149, 2012 Akashiba T, Kawahara S, Akahoshi T, et al. Relationship Between Quality of Life and Mood or Depression in Patients With Severe Obstructive Sleep Apnea Syndrome. CHEST 122: 861-865, 2002 Glebocka A, Kossowska A, Bednarek M. Obstructive sleep apnea and the quality of life. Journal of Physiology and Pharmacology 57: 111-117, 2006 Diamanti C, Manali E, Ginieri-Coccossis M, et al. Depression, physical activity, energy consumption, and quality of life in OSA patients before and after CPAP treatment. Sleep Breath 17(4):1159-68, 2013 Gagnadoux F, Le Vaillant M, Goupil F, et al. Depressive symptoms before and after long-term continuous positive airway pressure therapy in sleep apnea patients. CHEST 145(5):1025-1031, 2014